CLINICAL TRIAL: NCT01524991
Title: Phase II Trial of Gemcitabine, Cisplatin, Plus Ipilimumab as First-line Treatment for Patients With Metastatic Urothelial Carcinoma: Hoosier Cancer Research Network GU10-148
Brief Title: First-Line Gemcitabine, Cisplatin + Ipilimumab for Metastatic Urothelial Carcinoma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Hoosier Cancer Research Network (Other)
Collaborators: Bristol-Myers Squibb (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: GU10-148
Record Dates: First submitted 2012-01-30; First posted 2012-02-02 (Estimated); Results first posted 2019-11-29 (Actual); Last update posted 2022-07-11 (Actual); Status verified 2022-07

CONDITIONS: Urothelial Carcinoma
MeSH Terms: conditions — Carcinoma, Transitional Cell | interventions — Gemcitabine; Cisplatin; Ipilimumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Treatment (Experimental): Gemcitabine 1000 mg/m2 Days 1 & 8 Cisplatin 70 mg/m2 Day 1 Ipilimumab 10 mg/kg Day 1 (start cycle 3)
  Interventions: Drug: Gemcitabine; Drug: Cisplatin; Drug: Ipilimumab

INTERVENTIONS:
Drug: Gemcitabine — Gemcitabine 1000 mg/m2 Days 1 & 8 (all cycles)
Drug: Cisplatin — Cisplatin 70 mg/m2 Day 1 (all cycles)
Drug: Ipilimumab — Ipilimumab 10 mg/kg Day 1 (start cycle 3)

SUMMARY:
Gemcitabine plus cisplatin is standard treatment for advanced urothelial cancer. Ipilimumab has shown intriguing activity as neoadjuvant therapy in patients with clinically localized bladder cancer undergoing radical cystectomy. The combination of gemcitabine, cisplatin, plus ipilimumab may build on the chemosensitivity of urothelial carcinoma to produce more durable responses and improved outcomes.

DETAILED DESCRIPTION:
OUTLINE: This is a multi-center study

Gemcitabine 1000 mg/m2 Days 1 & 8 Cisplatin 70 mg/m2 Day 1 Ipilimumab 10 mg/kg Day 1 (start cycle 3)

Treatment during the induction phase will be administered in six 21-day cycles. During cycles 1 and 2, gemcitabine plus cisplatin will be administered WITHOUT ipilimumab. During cycles 3-6, combination therapy with gemcitabine, cisplatin, plus ipilimumab will be administered. Patients without evidence of disease progression (by irRC) after completion cycle 6 will continue single-agent ipilimumab maintenance every 3 months.

Karnofsky performance status (KPS) ≥ 80% within 14 days prior to registration for protocol therapy.

Life Expectancy: Not Specified

Hematopoietic:

* White blood cell count (WBC) ≥ 3.5K/mm3
* Hemoglobin (Hgb) ≥ 9 g/dL
* Platelets ≥ 100K/mm3
* Absolute neutrophil count (ANC) ≥ 1.5k/mm3

Hepatic:

* Bilirubin ≤ 1.5 times x Upper Limit of Normal (ULN) (except patients with Gilbert's Syndrome, who must have a total bilirubin less than 3.0 mg/dL)
* Aspartate aminotransferase (AST, SGOT) ≤ 2.5 x ULN. NOTE: If the patient has liver metastases present, then ≤ 5 x ULN

Renal:

* Calculated creatinine clearance of ≥ 55 cc/min using the Cockcroft-Gault formula

Cardiovascular: Not Specified

ELIGIBILITY:
Inclusion Criteria:

* Histological or cytological proof of urothelial carcinoma of the urethra, bladder, ureters, or renal pelvis.
* Advanced (clinical stage T4b, unresectable) or metastatic disease.
* Prior radiation therapy is allowed to < 25% of the bone marrow.
* Age > 18 years at the time of consent.
* Written informed consent and HIPAA authorization for release of personal health information.
* Females must not be pregnant or breastfeeding.
* WOCBP must have a negative serum or urine pregnancy test (minimum sensitivity 25 IU/L or equivalent units of HCG) within 72 hours before the start of ipilimumab.
* Men of fathering potential must be using an adequate method of contraception to avoid conception throughout the study [and for up to 26 weeks after the last dose of investigational product] in such a manner that the risk of pregnancy is minimized.
* Prior Autoimmune disease: Patients with a history of inflammatory bowel disease, including ulcerative colitis and Crohn's Disease, are excluded from this study, as are patients with a history of symptomatic disease (eg, rheumatoid arthritis, systemic progressive sclerosis [scleroderma], systemic lupus erythematosus, autoimmune vasculitis [eg, Wegener's Granulomatosis]); motor neuropathy considered of autoimmune origin (e.g. Guillain-Barre Syndrome and Myasthenia Gravis). Patients with other immune disorders should not be enrolled without discussion with the principal investigator.

Exclusion Criteria:

* No active CNS metastases. Subjects with neurological symptoms must undergo a head CT scan or brain MRI to exclude brain metastasis.
* No prior malignancy is allowed except for cancers that have been definitively treated with a risk of recurrence of < 30% based on the treating oncologists assessment.
* Patients may not have received prior systemic chemotherapy for metastatic/advanced urothelial carcinoma. Prior neoadjuvant/adjuvant therapy is permitted if completed ≥ 12 months prior to registration for protocol therapy. Prior intravesical therapy is permitted.
* No treatment with any investigational agent within 30 days prior to registration for protocol therapy.
* No underlying medical or psychiatric condition, which in the opinion of the investigator will make the administration of ipilimumab hazardous or obscure the interpretation of AEs, such as a condition associated with frequent diarrhea.
* No non-oncology vaccine therapy used for prevention of infectious diseases (for up to 1 month before or after any dose of ipilimumab).
* No history of prior treatment with ipilimumab or prior CD137 agonist or CTLA 4 inhibitor or agonist.
* No known active or chronic infection with HIV, Hepatitis B, or Hepatitis C.
* No clinically significant infections as judged by the treating investigator.
* No chronic systemic corticosteroids (defined as the equivalent of prednisone ≥ 20 mg PO daily for > 6 months during the past year)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Actual)
Dates: Start 2012-01 (Actual); Primary Completion 2017-07-15 (Actual); Study Completion 2018-12-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Matthew Galsky, M.D., Study Chair — Hoosier Cancer Research Network
Locations (8):
- United States (8):
  - City of Hope: Duarte, Duarte, California
  - IU Health Goshen Hospital, Goshen, Indiana
  - Indiana University Melvin & Bren Simon Cancer Center, Indianapolis, Indiana
  - IU Health Central Indiana Cancer Centers, Indianapolis, Indiana
  - Nebraska Cancer Specialists, Omaha, Nebraska
  - Tisch Cancer Institute at Mount Sinai Medical Center, New York, New York
  - Texas Oncology, PA, Dallas, Texas
  - Virginia Oncology Associates, Norfolk, Virginia

REFERENCES:
- [Background] Galsky MD, Hahn NM, Albany C, Fleming MT, Starodub A, Twardowski P, Hauke RJ, Sonpavde G, Merad M, Gnjatic S, Bhardwaj N, Chippada-Venkata U, Oh WK, Kim-Schulze S. Impact of gemcitabine + cisplatin + ipilimumab on circulating immune cells in patients (pts) with metastatic urothelial cancer (mUC). J Clin Oncol 33:5s, 2015 (suppl; abstr 4586)
- [Derived] Galsky MD, Wang H, Hahn NM, Twardowski P, Pal SK, Albany C, Fleming MT, Starodub A, Hauke RJ, Yu M, Zhao Q, Sonpavde G, Donovan MJ, Patel VG, Sfakianos JP, Domingo-Domenech J, Oh WK, Akers N, Losic B, Gnjatic S, Schadt EE, Chen R, Kim-Schulze S, Bhardwaj N, Uzilov AV. Phase 2 Trial of Gemcitabine, Cisplatin, plus Ipilimumab in Patients with Metastatic Urothelial Cancer and Impact of DNA Damage Response Gene Mutations on Outcomes. Eur Urol. 2018 May;73(5):751-759. doi: 10.1016/j.eururo.2017.12.001. Epub 2017 Dec 13. PMID 29248319
- See also: Hoosier Cancer Research Network Homepage — http://www.hoosiercancer.org

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Treatment
Started | 36
Completed | 2
Not Completed | 34
Not completed — Adverse Event | 12
Not completed — Death | 1
Not completed — Disease ProgressionDu | 17
Not completed — Other complicating disease | 1
Not completed — Withdrawal by Subject | 2
Not completed — Symptomatic Deterioration | 1

BASELINE CHARACTERISTICS:
Arm/Group | Treatment
Number analyzed (Participants) | 36
Age, Continuous [Median (Full Range); unit: years] | 36 [33 to 80]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7
  Male | 29
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 4
  Not Hispanic or Latino | 32
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 1
  White | 35
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 36
Karnovsky Performance Status [Count of Participants; unit: Participants] — Karnofsky Performance Status (KPS) is a general indicator of a subject's well being and ability to carry on daily activities. The KPS scale ranges from 0-100 in 10 unit increments where 100=Normal; no complaints; no evidence of disease and 0=Dead
  Participants
    KPS 100 | 9
    KPS 90 | 16
    KPS 80 | 11

OUTCOME MEASURES:

1. Primary Outcome: Median Overall Survival
Description: To determine the median overall survival of patients with advanced/metastatic urothelial cancer treated with gemcitabine, cisplatin, plus ipilimumab, calculated from the date of registration until the date of final analysis, projected to be 48 months from the start of the study.
Time Frame: 48 months
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Treatment
Number analyzed (Participants) | 36
months | 13.9 [10.5 to 23.4]

2. Secondary Outcome: Progression-Free Survival
Description: To determine the progression-free survival (using irRC and RECIST v1.0) of patients with advanced/metastatic urothelial carcinoma treated with gemcitabine, cisplatin, and ipilimumab.
  Progression is defined using Response Evaluation Criteria In Solid Tumors Criteria (RECIST v1.0), as a 20% increase in the sum of the longest diameter of target lesions, or a measurable increase in a non-target lesion, or the appearance of new lesions". Progression is definied by IrRC as "at least 25% increase in tumor burden compared with nadir (at any single time point) in two consecutive observations at least 4 wk apart."
Time Frame: 12 months
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Treatment
Number analyzed (Participants) | 36
months | 7.9 [6.4 to 9.9]

3. Secondary Outcome: Best Overall Response Rate
Description: To determine the best overall response rate to treatment with gemcitabine, cisplatin, plus ipilimumab, per RECIST 1.1 criteria.
Time Frame: 12 months
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment
Number analyzed (Participants) | 36
Participants
  Complete Response (CR) | 6
  Partial Response (PR) | 19
  Stable Disease (SD) | 10
  Progressive Disease (PD) | 1

4. Secondary Outcome: Number of Adverse Events Experienced by Patients
Description: To determine the safety of treatment with gemcitabine, cisplatin, plus ipilimumab. The highest grade adverse event for each subject is presented.
Time Frame: 12 months
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment
Number analyzed (Participants) | 36
Participants
  Grade 1 | 1
  Grade 2 | 6
  Grade 3 | 19
  Grade 4 | 10

ADVERSE EVENTS:
Time Frame: From the start of treatment to 30 days following the last treatment, a maximum of 1 year
Arm/Group | Treatment
All-Cause Mortality (participants affected / at risk) | 28/36
Serious Adverse Events (participants affected / at risk) | 18/36
Other Adverse Events (participants affected / at risk) | 36/36
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Treatment (N=36)
ACUTE KIDNEY INJURY (Renal and urinary disorders) | 3 (3)
ADRENAL INSUFFICIENCY (Endocrine disorders) | 1 (1)
ANEMIA (Blood and lymphatic system disorders) | 1 (1)
ATRIAL FIBRILLATION (Cardiac disorders) | 2 (2)
AUTOIMMUNE DISORDER (Immune system disorders) | 2 (3)
COLITIS (Gastrointestinal disorders) | 1 (2)
CREATININE INCREASED (Investigations) | 1 (1)
DIARRHEA (Gastrointestinal disorders) | 2 (3)
ENDOCRINE DISORDERS - OTHER, SPECIFY (Endocrine disorders) | 1 (1)
FEVER (General disorders) | 4 (5)
HYPERTHYROIDISM (Endocrine disorders) | 1 (1)
HYPONATREMIA (Metabolism and nutrition disorders) | 1 (2)
LUNG INFECTION (Infections and infestations) | 1 (1)
OBSTRUCTION GASTRIC (Gastrointestinal disorders) | 1 (1)
PERIPHERAL MOTOR NEUROPATHY (Nervous system disorders) | 1 (1)
RECTAL PAIN (Gastrointestinal disorders) | 1 (1)
SEPSIS (Infections and infestations) | 1 (1)
SMALL INTESTINAL OBSTRUCTION (Gastrointestinal disorders) | 1 (2)
THROMBOEMBOLIC EVENT (Vascular disorders) | 5 (9)
UPPER GASTROINTESTINAL HEMORRHAGE (Gastrointestinal disorders) | 1 (1)
UPPER RESPIRATORY INFECTION (Infections and infestations) | 1 (1)
URINARY TRACT INFECTION (Infections and infestations) | 3 (3)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Treatment (N=36)
ABDOMINAL DISTENSION (Gastrointestinal disorders) | 1 (1)
ABDOMINAL PAIN (Gastrointestinal disorders) | 14 (19)
ADRENAL INSUFFICIENCY (Endocrine disorders) | 2 (2)
AGITATION (Psychiatric disorders) | 2 (2)
ALANINE AMINOTRANSFERASE INCREASED (Investigations) | 5 (7)
ALKALINE PHOSPHATASE INCREASED (Investigations) | 5 (10)
ALLERGIC REACTION (Immune system disorders) | 1 (1)
ALLERGIC RHINITIS (Respiratory, thoracic and mediastinal disorders) | 4 (4)
ALOPECIA (Skin and subcutaneous tissue disorders) | 10 (12)
ANEMIA (Blood and lymphatic system disorders) | 24 (109)
ANOREXIA (Metabolism and nutrition disorders) | 19 (30)
ANXIETY (Psychiatric disorders) | 7 (7)
ARTHRALGIA (Musculoskeletal and connective tissue disorders) | 4 (4)
ARTHRITIS (Musculoskeletal and connective tissue disorders) | 1 (1)
ASCITES (Gastrointestinal disorders) | 1 (1)
ASPARTATE AMINOTRANSFERASE INCREASED (Investigations) | 4 (7)
ATRIAL FIBRILLATION (Cardiac disorders) | 3 (4)
BACK PAIN (Musculoskeletal and connective tissue disorders) | 11 (17)
BLADDER SPASM (Renal and urinary disorders) | 1 (1)
BLOATING (Gastrointestinal disorders) | 1 (1)
BLOOD BILIRUBIN INCREASED (Investigations) | 1 (1)
BLURRED VISION (Eye disorders) | 4 (4)
BONE PAIN (Musculoskeletal and connective tissue disorders) | 4 (4)
BRUISING (Injury, poisoning and procedural complications) | 1 (1)
CATARACT (Eye disorders) | 1 (1)
CHEST PAIN - CARDIAC (Cardiac disorders) | 1 (1)
CHEST WALL PAIN (Musculoskeletal and connective tissue disorders) | 1 (1)
CHILLS (General disorders) | 7 (9)
CHOLESTEROL HIGH (Investigations) | 4 (4)
COLITIS (Gastrointestinal disorders) | 4 (4)
CONSTIPATION (Gastrointestinal disorders) | 24 (34)
COUGH (Respiratory, thoracic and mediastinal disorders) | 18 (24)
CREATININE INCREASED (Investigations) | 12 (26)
DEHYDRATION (Metabolism and nutrition disorders) | 7 (11)
DELIRIUM (Psychiatric disorders) | 2 (2)
DEPRESSION (Psychiatric disorders) | 6 (6)
DIARRHEA (Gastrointestinal disorders) | 23 (40)
DIZZINESS (Nervous system disorders) | 11 (14)
DRY SKIN (Skin and subcutaneous tissue disorders) | 4 (4)
DYSGEUSIA (Nervous system disorders) | 11 (13)
DYSPEPSIA (Gastrointestinal disorders) | 9 (11)
DYSPHAGIA (Gastrointestinal disorders) | 1 (2)
DYSPNEA (Respiratory, thoracic and mediastinal disorders) | 16 (18)
EAR PAIN (Ear and labyrinth disorders) | 1 (1)
EDEMA LIMBS (General disorders) | 11 (15)
ENCEPHALOPATHY (Nervous system disorders) | 1 (1)
ENDOCRINE DISORDERS - OTHER, SPECIFY (Endocrine disorders) | 4 (5)
EPISTAXIS (Respiratory, thoracic and mediastinal disorders) | 2 (4)
ERECTILE DYSFUNCTION (Reproductive system and breast disorders) | 1 (1)
ERYTHEMA MULTIFORME (Skin and subcutaneous tissue disorders) | 1 (1)
FALL (Injury, poisoning and procedural complications) | 1 (1)
FATIGUE (General disorders) | 33 (71)
FEVER (General disorders) | 12 (17)
FLANK PAIN (Musculoskeletal and connective tissue disorders) | 6 (8)
FLU LIKE SYMPTOMS (General disorders) | 2 (2)
GAIT DISTURBANCE (General disorders) | 1 (1)
GASTROESOPHAGEAL REFLUX DISEASE (Gastrointestinal disorders) | 5 (5)
GASTROINTESTINAL DISORDERS - OTHER, SPECIFY (Gastrointestinal disorders) | 2 (2)
GASTROINTESTINAL PAIN (Gastrointestinal disorders) | 1 (1)
GENERAL DISORDERS AND ADMINISTRATION SITE CONDITIONS - OTHER, SPECIFY (General disorders) | 2 (2)
GENERALIZED MUSCLE WEAKNESS (Musculoskeletal and connective tissue disorders) | 4 (5)
GENITAL EDEMA (Reproductive system and breast disorders) | 2 (2)
HEADACHE (Nervous system disorders) | 12 (17)
HEARING IMPAIRED (Ear and labyrinth disorders) | 1 (1)
HEMATURIA (Renal and urinary disorders) | 10 (11)
HICCUPS (Respiratory, thoracic and mediastinal disorders) | 5 (5)
HOARSENESS (Respiratory, thoracic and mediastinal disorders) | 1 (1)
HOT FLASHES (Vascular disorders) | 1 (1)
HYPERCALCEMIA (Metabolism and nutrition disorders) | 1 (2)
HYPERGLYCEMIA (Metabolism and nutrition disorders) | 6 (9)
HYPERHIDROSIS (Skin and subcutaneous tissue disorders) | 1 (1)
HYPERKALEMIA (Metabolism and nutrition disorders) | 4 (9)
HYPERTENSION (Vascular disorders) | 10 (11)
HYPERTHYROIDISM (Endocrine disorders) | 2 (2)
HYPERTRIGLYCERIDEMIA (Metabolism and nutrition disorders) | 2 (2)
HYPERURICEMIA (Metabolism and nutrition disorders) | 1 (1)
HYPOALBUMINEMIA (Metabolism and nutrition disorders) | 5 (18)
HYPOCALCEMIA (Metabolism and nutrition disorders) | 3 (3)
HYPOGLYCEMIA (Metabolism and nutrition disorders) | 1 (2)
HYPOKALEMIA (Metabolism and nutrition disorders) | 9 (19)
HYPOMAGNESEMIA (Metabolism and nutrition disorders) | 9 (26)
HYPONATREMIA (Metabolism and nutrition disorders) | 17 (41)
HYPOPHOSPHATEMIA (Metabolism and nutrition disorders) | 3 (3)
HYPOTENSION (Vascular disorders) | 2 (3)
HYPOTHYROIDISM (Endocrine disorders) | 4 (5)
HYPOXIA (Respiratory, thoracic and mediastinal disorders) | 2 (2)
INFECTIONS AND INFESTATIONS - OTHER, SPECIFY (Infections and infestations) | 4 (5)
INJURY, POISONING AND PROCEDURAL COMPLICATIONS - OTHER, SPECIFY (Injury, poisoning and procedural complications) | 1 (3)
INSOMNIA (Psychiatric disorders) | 11 (12)
INVESTIGATIONS - OTHER, SPECIFY (Investigations) | 1 (1)
KIDNEY INFECTION (Infections and infestations) | 1 (1)
LEUKOCYTOSIS (Blood and lymphatic system disorders) | 1 (1)
LIP INFECTION (Infections and infestations) | 1 (1)
LOCALIZED EDEMA (General disorders) | 1 (1)
LYMPHEDEMA (Vascular disorders) | 1 (1)
LYMPHOCYTE COUNT DECREASED (Investigations) | 5 (13)
MALAISE (General disorders) | 1 (1)
MEMORY IMPAIRMENT (Nervous system disorders) | 1 (1)
METABOLISM AND NUTRITION DISORDERS - OTHER, SPECIFY (Metabolism and nutrition disorders) | 1 (1)
MUCOSITIS ORAL (Gastrointestinal disorders) | 4 (6)
MUSCLE WEAKNESS UPPER LIMB (Musculoskeletal and connective tissue disorders) | 1 (1)
MYALGIA (Musculoskeletal and connective tissue disorders) | 1 (1)
NASAL CONGESTION (Respiratory, thoracic and mediastinal disorders) | 3 (3)
NAUSEA (Gastrointestinal disorders) | 27 (64)
NECK PAIN (Musculoskeletal and connective tissue disorders) | 1 (1)
NEOPLASMS BENIGN, MALIGNANT AND UNSPECIFIED (INCL CYSTS AND POLYPS) - OTHER, SPECIFY (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
NERVOUS SYSTEM DISORDERS - OTHER, SPECIFY (Nervous system disorders) | 1 (1)
NEURALGIA (Nervous system disorders) | 1 (1)
NEUTROPHIL COUNT DECREASED (Investigations) | 21 (56)
NON-CARDIAC CHEST PAIN (General disorders) | 2 (2)
OBESITY (Metabolism and nutrition disorders) | 1 (1)
OBSTRUCTION GASTRIC (Gastrointestinal disorders) | 1 (1)
ORAL PAIN (Gastrointestinal disorders) | 1 (1)
PAIN (General disorders) | 15 (22)
PAIN IN EXTREMITY (Musculoskeletal and connective tissue disorders) | 10 (15)
PAIN OF SKIN (Skin and subcutaneous tissue disorders) | 1 (1)
PALPITATIONS (Cardiac disorders) | 2 (2)
PAPULOPUSTULAR RASH (Infections and infestations) | 1 (1)
PARESTHESIA (Nervous system disorders) | 2 (2)
PELVIC PAIN (Reproductive system and breast disorders) | 3 (3)
PERIPHERAL MOTOR NEUROPATHY (Nervous system disorders) | 1 (1)
PERIPHERAL SENSORY NEUROPATHY (Nervous system disorders) | 16 (20)
PHLEBITIS (Vascular disorders) | 1 (1)
PLATELET COUNT DECREASED (Investigations) | 17 (38)
PNEUMONITIS (Respiratory, thoracic and mediastinal disorders) | 2 (2)
PRODUCTIVE COUGH (Respiratory, thoracic and mediastinal disorders) | 1 (2)
PROSTATIC OBSTRUCTION (Reproductive system and breast disorders) | 1 (1)
PROTEINURIA (Renal and urinary disorders) | 1 (1)
PRURITUS (Skin and subcutaneous tissue disorders) | 7 (9)
PULMONARY EDEMA (Respiratory, thoracic and mediastinal disorders) | 2 (2)
PULMONARY FIBROSIS (Respiratory, thoracic and mediastinal disorders) | 1 (1)
PURPURA (Skin and subcutaneous tissue disorders) | 1 (1)
RASH ACNEIFORM (Skin and subcutaneous tissue disorders) | 7 (9)
RASH MACULO-PAPULAR (Skin and subcutaneous tissue disorders) | 7 (13)
RASH PUSTULAR (Infections and infestations) | 1 (1)
RECTAL HEMORRHAGE (Gastrointestinal disorders) | 2 (2)
RECTAL PAIN (Gastrointestinal disorders) | 1 (2)
RENAL AND URINARY DISORDERS - OTHER, SPECIFY (Renal and urinary disorders) | 7 (9)
RENAL CALCULI (Renal and urinary disorders) | 1 (1)
RESPIRATORY FAILURE (Respiratory, thoracic and mediastinal disorders) | 1 (1)
RESPIRATORY, THORACIC AND MEDIASTINAL DISORDERS - OTHER, SPECIFY (Respiratory, thoracic and mediastinal disorders) | 1 (1)
RESTLESSNESS (Psychiatric disorders) | 1 (1)
SINUS BRADYCARDIA (Cardiac disorders) | 1 (1)
SINUS DISORDER (Respiratory, thoracic and mediastinal disorders) | 1 (1)
SINUS TACHYCARDIA (Cardiac disorders) | 1 (1)
SKIN AND SUBCUTANEOUS TISSUE DISORDERS - OTHER, SPECIFY (Skin and subcutaneous tissue disorders) | 6 (6)
SKIN INFECTION (Infections and infestations) | 5 (7)
SKIN ULCERATION (Skin and subcutaneous tissue disorders) | 1 (1)
SMALL INTESTINAL OBSTRUCTION (Gastrointestinal disorders) | 1 (1)
SMALL INTESTINE INFECTION (Infections and infestations) | 1 (1)
SNEEZING (Respiratory, thoracic and mediastinal disorders) | 2 (3)
SOMNOLENCE (Nervous system disorders) | 1 (1)
SORE THROAT (Respiratory, thoracic and mediastinal disorders) | 3 (6)
SUPERFICIAL THROMBOPHLEBITIS (Vascular disorders) | 2 (2)
SURGICAL AND MEDICAL PROCEDURES - OTHER, SPECIFY (Surgical and medical procedures) | 2 (2)
SYNCOPE (Nervous system disorders) | 1 (1)
THROMBOEMBOLIC EVENT (Vascular disorders) | 6 (7)
TINNITUS (Ear and labyrinth disorders) | 4 (7)
TREMOR (Nervous system disorders) | 3 (3)
UPPER RESPIRATORY INFECTION (Infections and infestations) | 1 (1)
URINARY FREQUENCY (Renal and urinary disorders) | 6 (7)
URINARY INCONTINENCE (Renal and urinary disorders) | 2 (2)
URINARY RETENTION (Renal and urinary disorders) | 2 (2)
URINARY TRACT INFECTION (Infections and infestations) | 11 (14)
URINARY TRACT PAIN (Renal and urinary disorders) | 1 (1)
URINARY URGENCY (Renal and urinary disorders) | 1 (1)
VASCULAR DISORDERS - OTHER, SPECIFY (Vascular disorders) | 1 (1)
VOMITING (Gastrointestinal disorders) | 14 (35)
WEIGHT GAIN (Investigations) | 2 (9)
WEIGHT LOSS (Investigations) | 7 (12)
WHITE BLOOD CELL DECREASED (Investigations) | 7 (18)
WOUND INFECTION (Infections and infestations) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2014-05-22): https://cdn.clinicaltrials.gov/large-docs/91/NCT01524991/Prot_SAP_000.pdf